CLINICAL TRIAL: NCT01833754
Title: A Phase 1, Open-label, Single-dose Study of Romosozumab (AMG 785) Administered Subcutaneously to Healthy Subjects and Subjects With Stage 4 Renal Impairment or Stage 5 Renal Impairment Requiring Hemodialysis
Brief Title: Study of Romosozumab (AMG 785) Administered to Healthy Participants and Patients With Stage 4 Renal Impairment or Stage 5 Renal Impairment Requiring Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110227
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, Bone, Renal, Insufficiency, Kidney, Hemodialysis, Impairment
MeSH Terms: conditions — Osteoporosis | interventions — romosozumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Stage 4 Renal Impairment (Experimental): Participants with stage 4 renal impairment (defined as an estimated glomerular filtration rate [eGFR] 15 to 29 mL/min/1.73 m²) received a single subcutaneous injection of 210 mg romosozumab on day 1.
  Interventions: Drug: Romosozumab
- Group 2: ESRD Requiring Hemodialysis (Experimental): Participants with end stage renal disease (ESRD) requiring hemodialysis received a single subcutaneous injection of 210 mg romosozumab on day 1.
  Interventions: Drug: Romosozumab
- Group 3: Healthy Participants (Experimental): Healthy participants (eGFR ≥ 80 mL/min/1.73 m²) received a single subcutaneous injection of 210 mg romosozumab on day 1.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered as three 70 mg/mL prefilled syringe injections
  Other Names: AMG 785; EVENITY™

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity profile of romosozumab after a single 210 mg subcutaneous dose in healthy participants and patients with stage 4 renal impairment (RI) or stage 5 RI requiring hemodialysis.

ELIGIBILITY:
INCLUSION CRITERIA - ALL SUBJECTS :

* Males or females ≥ 50 years of age
* Body weight ≥ 45 and ≤ 110 kg
* Willing to adhere to calcium and vitamin D supplementation requirements
* Females must be of non-reproductive potential

INCLUSION CRITERIA - SUBJECTS WITH RENAL IMPAIRMENT (GROUPS 1 AND 2):

* Group 1 - Stage 4 RI (estimated glomerular filtration rate (eGFR) 15-29 mL/min/1.73 m²)
* Group 2 - End stage renal disease requiring hemodialysis

INCLUSION CRITERIA - HEALTHY SUBJECTS (GROUP 3):

• Renal function defined as an estimated glomerular filtration rate (eGFR) ≥ 80 mL/min/1.73 m²

EXCLUSION CRITERIA - ALL SUBJECTS:

* History of metabolic or bone disease (except for metabolic bone disease in renal impairment (RI) subjects)
* History of osteoporosis, vertebral fracture, or fragility fracture of the wrist, humerus, hip, or pelvis after age 50
* Recent bone fracture
* Vitamin D insufficiency
* Hypocalcemia or hypercalcemia
* Hypomagnesemia
* Hypophosphatemia
* Untreated hyper- or hypothyroidism
* Females with a positive pregnancy test
* Males with pregnant partners
* Females who are lactating/breastfeeding or plan to breastfeed on study and for 3 months after receiving the dose of study drug
* History of spinal stenosis
* History of facial nerve paralysis
* Positive for human immunodeficiency virus (HIV) antibodies
* Positive for hepatitis B surface antigen or detectable hepatitis C
* Malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical, or breast ductal carcinoma in situ) within 5 years before screening
* History of solid organ or bone marrow transplants EXCLUSION CRITERIA - HEALTHY SUBJECTS (GROUP 3)
* Current hyper- or hypoparathyroidism

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2014-02-19 (Actual); Study Completion 2014-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Research Site, Tempe, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Pembroke Pines, Florida
  - Research Site, Orangeburg, South Carolina

REFERENCES:
- [Background] Hsu CP, Maddox J, Block G, Bartley Y, Yu Z. Influence of Renal Function on Pharmacokinetics, Pharmacodynamics, and Safety of a Single Dose of Romosozumab. J Clin Pharmacol. 2022 Sep;62(9):1132-1141. doi: 10.1002/jcph.2050. Epub 2022 Apr 2. PMID 35304747
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in the United States. The first participant enrolled on 22 April 2013 and the last participant enrolled on 05 November 2013.
Period: Overall Study
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.4) | 65.1 (6.7) | 63.0 (8.8) | 64.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7 | 14
  Male | 4 | 5 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 10
  Not Hispanic or Latino | 4 | 4 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Black or African American | 1 | 3 | 1 | 5
  White | 6 | 5 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event was defined as an adverse event (AE) that met at least 1 of the following serious criteria:
  * fatal
  * life-threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. A treatment-related adverse event (TRAE) was an AE assessed by the investigator as possibly related to the study drug, indicated by a "yes" response to the question: "Is there a reasonable possibility that the event may have been caused by the investigational product?"
Time Frame: From the first dose of study drug up to day 85
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
Participants
  All adverse events | 7 | 6 | 0
  Serious adverse events | 1 | 1 | 0
  AEs leading to discontinuation of study drug | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0
  Treatment-related adverse events | 5 | 6 | 0
  Treatment-related serious adverse events | 0 | 0 | 0
  TRAEs leading to discontinuation of study drug | 0 | 0 | 0
  Treatment-related fatal adverse events | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Romosozumab
Time Frame: Pre-dose on day -1 and on days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 36, 43, 57 and 85
Population: All participants were included in the analysis
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µg/mL | 28.9 (10.8) | 19.8 (7.3) | 22.4 (10.3)

3. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) of Romosozumab
Time Frame: Pre-dose on day -1 and on days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 36, 43, 57 and 85
Population: All participants were included in the analysis
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
days | 5.0 (10.8) [3.0 to 7.0] | 5.0 (7.3) [3.0 to 7.0] | 5.0 (10.3) [3.0 to 7.0]

4. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Time Frame: Pre-dose on day -1 and on days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 36, 43, 57 and 85
Population: All participants were included in the analysis
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
days*µg/mL | 637 (218) | 444 (154) | 443 (143)

5. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Time Frame: Pre-dose on day -1 and on days 2, 3, 4, 6, 8, 11, 15, 18, 22, 29, 36, 43, 57 and 85
Population: All participants were included in the analysis
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
days*µg/mL | 642 (221) | 447 (154) | 445 (143)

6. Primary Outcome: Number of Participants Who Developed Anti-Romosozumab Antibodies
Description: Two validated assays were used to detect the presence of anti-romosozumab antibodies. First, an electrochemiluminescent immunoassay was used to detect binding antibodies (screening assay) and confirm antibodies (confirmatory assay) capable of binding romosozumab. Second, a non-cell-based competitive binding bioassay was used to test positive binding antibody samples for neutralizing activity against romosozumab.
  If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the participant was defined as positive for neutralizing antibodies.
Time Frame: Baseline and day 85
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Binding antibody positive | 0 | 0 | 1
  Neutralizing antibody positive | 0 | 0 | 0

7. Primary Outcome: Albumin-Adjusted Serum Calcium Concentrations by Visit
Description: Albumin-adjusted calcium was derived as:
  Where serum albumin < 40 g/L then albumin-adjusted calcium = measured total calcium (mmol/L) + 0.02 * [40 - serum albumin (g/L)]; Where serum albumin ≥ 40 g/L then albumin-adjusted calcium = measured total calcium.
Time Frame: Baseline, days 8, 15, 22, 29, 43, 57, and 85/end of study visit
Population: All participants who received study drug
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
mmol/L
  Baseline | 2.452 (0.228) | 2.379 (0.131) | 2.340 (0.057)
  Day 8 | 2.355 (0.187) | 2.226 (0.205) | 2.308 (0.072)
  Day 15 | 2.378 (0.146) | 2.194 (0.107) | 2.293 (0.070)
  Day 22 | 2.329 (0.151) | 2.074 (0.193) | 2.311 (0.104)
  Day 29 | 2.338 (0.162) | 2.166 (0.258) | 2.316 (0.062)
  Day 43 | 2.404 (0.200) | 2.209 (0.169) | 2.320 (0.065)
  Day 57 | 2.406 (0.179) | 2.284 (0.114) | 2.319 (0.070)
  End of Study | 2.428 (0.201) | 2.291 (0.264) | 2.330 (0.065)

8. Primary Outcome: Intact Parathyroid Hormone (iPTH)Concentrations by Visit
Time Frame: Baseline, days 8, 15, 22, 29, 43, 57, and 85/end of study visit
Population: All participants who received study drug and with available data at each time point
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
pmol/L
  Baseline | 5.014 (1.597) | 11.765 (12.003) | 4.682 (3.432)
  Day 8: number analyzed (Participants) | 8 | 7 | 7
  Day 8 | 9.192 (3.077) | 19.812 (16.289) | 6.776 (3.612)
  Day 15 | 8.887 (4.743) | 17.376 (10.108) | 6.473 (3.880)
  Day 22 | 10.425 (4.190) | 29.724 (20.565) | 6.818 (3.959)
  Day 29 | 12.495 (5.248) | 29.857 (20.461) | 7.348 (3.997)
  Day 43: number analyzed (Participants) | 8 | 7 | 6
  Day 43 | 9.921 (5.906) | 21.374 (14.184) | 6.508 (3.289)
  Day 57 | 9.311 (4.571) | 17.893 (11.196) | 5.279 (2.215)
  End of Study: number analyzed (Participants) | 7 | 8 | 8
  End of Study | 6.958 (3.812) | 23.503 (24.339) | 4.457 (2.506)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to day 85.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Group 1: Stage 4 Renal Impairment | Group 2: ESRD Requiring Hemodialysis | Group 3: Healthy Participants
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 6/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Stage 4 Renal Impairment (N=8) | Group 2: ESRD Requiring Hemodialysis (N=8) | Group 3: Healthy Participants (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Stage 4 Renal Impairment (N=8) | Group 2: ESRD Requiring Hemodialysis (N=8) | Group 3: Healthy Participants (N=8)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 4 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.